CLINICAL TRIAL: NCT04007094
Title: A Prospective, Single Arm Study of Patients Undergoing Posterolateral Lumbar Fusion (Without Interbody) Supplemented With ViviGen Cellular Bone Matrix
Brief Title: Single-Armed Use of ViviGen Cellular Bone Matrix in Patients Undergoing Posterolateral Lumbar Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary Investigator left university. Site completing follow up assessments for previously enrolled subject only.
Sponsor: Ohio State University (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Principal Investigator, Andrew Grossbach, Assistant Professor, Department of Neurological Surgery, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018H0253
Record Dates: First submitted 2019-04-24; First posted 2019-07-05 (Actual); Results first posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-05

CONDITIONS: Degenerative Disc Disease; Spinal Stenosis; Spondylosis; Spondylolisthesis
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis; Spondylosis; Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Arm (Experimental): Participants will be entered into the single armed study in which one side of the fusion will be coated with milled local autograft bone and the opposite fusion side will be supplemented with an equal volume of Depuy Synthes ViviGen.
  Interventions: Other: ViviGen Cellular Bone Matrix

INTERVENTIONS:
Other: ViviGen Cellular Bone Matrix — ViviGen Cellular Bone Matrix is a formulation of cryopreserved viable cortical cancellous bone matrix and demineralized bone. ViviGen is a Human Cells, Tissues, and Cellular and Tissue-based Product (HCT/P) as defined by the U.S. Food and Drug Administration in 21 CFR 1271.10

SUMMARY:
This is a prospective, single-arm post market study of patients to assess fusion in one or multiple continuous levels of the lumbosacral spine (L1-S1) using ViviGen Cellular Bone Matrix. All subjects will be followed out to 24 months for final assessment.

DETAILED DESCRIPTION:
Lumbar spine fusion rates can vary according to the surgical technique. Although many studies on spinal fusion have been conducted and reported, the heterogeneity of the study designs and data handling make it difficult to identify which approach yields the highest fusion rate. Traditional posterolateral intertransverse fusion (PLF) still remains a good procedure with acceptable fusion rates for most degenerative conditions. For solid fusion, PLF can be combined with interbody fusion to circumferentially stabilize the relevant segment, even though it is unclear whether this improves fusion rates.

A bone graft or bone graft substitute is required to produce the fusion and can be implanted on its own, in the posterolateral gutters, or contained with an interbody device using either a posterior or anterior approach. Spinal laminectomy is most often the largest generator of bone graft product due to the nature of the procedure. The current gold standard is autograft bone, in which tissue is harvested locally or from the iliac crest and is then placed at the site. However, local bone graft may be relatively limited and harvesting at the iliac crest can easily lead to significant morbidity. Complications such as inflammation, infection, and chronic pain may outlast the pain of the original surgical procedure.

Autograft is the gold standard because it possesses all of the characteristics necessary for new bone growth-namely, osteoconductivity, osteogenicity, and osteoinductivity. Allograft tissues are alternatives to autografts and are taken from donors or cadavers, circumventing some of the shortcomings of autografts by eliminating donor-site morbidity and issues of limited supply. Osteoconductivity refers to the situation in which the graft supports the attachment of new osteoblasts and osteoprogenitor cells, providing an interconnected structure through which new cells can migrate and new vessels can form. Osteogenicity refers to the situation when the osteoblasts that are at the site of new bone formation are able to produce minerals to calcify the collagen matrix that forms the substrate for new bone. Osteoinductivity refers to the ability of a graft to induce nondifferentiated stem cells or osteoprogenitor cells to differentiate into osteoblasts. Using the 2 basic criteria of a successful graft, osteoconduction and osteoinduction, investigators have developed several alternatives, some of which are available for clinical use and others of which are still in the developmental stage. Many of these alternatives use a variety of materials, including natural and synthetic polymers, ceramics, and composites, whereas others have incorporated factor- and cell-based strategies that are used either alone or in combination with other materials.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled to undergo a single or multilevel posterolateral spinal fusion surgery using ViviGen Cellular Bone matrix
* Subject must be over the age of 18 years old
* Subject has been unresponsive to conservative care for a minimum of 6 months.
* The subject must in the investigator's opinion, be psychosocially, mentally, and physically able to fully comply with this protocol including the required follow-up visits, the filling out of required forms, and have the ability to understand and give written informed consent.

Exclusion Criteria:

* Subjects requiring additional bone grafting materials other than local autograft and ViviGen Cellular Bone Matrix will be excluded from this outcomes study.
* Subject has inadequate tissue coverage over the operative site
* Subject has an open wound local to the operative area, or rapid joint disease, bone absorption, or osteoporosis.
* Subject has a condition requiring medications that may interfere with bone or soft tissue healing (i.e., oral or parenteral glucocorticoids, immunosuppressives, methotrexate, etc.).
* Subject has an active local or systemic infection.
* Subject has a metal sensitivity/foreign body sensitivity.
* Subject is morbidly obese, defined as a body mass index (BMI) greater than 45.
* Subject has any medical condition or extenuating circumstance that, in the opinion of the investigator, would preclude participation in the study.
* Subject is currently involved in another investigational drug or device study that could confound study data.
* Subject has a history (present or past) of substance abuse (recreational drugs, prescription drugs or alcohol) that in the investigator's opinion may interfere with protocol assessments and/or with the subject's ability to complete the protocol required follow-up.
* Subjects who are pregnant or plan to become pregnant in the next 24 months or who are lactating.
* Subject is involved in or planning to engage in litigation or receiving Worker's Compensation related to neck or back pain.
* Osteoporosis (per the investigator's diagnosis or per a T-score > 2.5 standard deviations below the mean for a young, healthy adult) that may prevent adequate fixation of screws and thus preclude the use of a pedicle screw system.
* Subjects who have a known or suspected allergy to any of the following antibiotics and/or reagents: Gentamicin Sulfate, Meropenem, Vancomycin, Dimethyl Sulfoxide (DMSO), and Human Serum Albumin (HSA);
* Immune compromised subjects
* Known sensitivity to device materials
* Subject is a prisoner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Vertebral Levels
Groups:
- Left Side - Local Autograft Bone: Left side fusion levels coated with milled local autograft bone
- Right Side - ViviGen: Right side Fusion Levels Supplemented with Depuy Synthes VigiGen
Period: Overall Study
Arm/Group | Left Side - Local Autograft Bone | Right Side - ViviGen
Started | 21; 58 Vertebral Levels | 21; 58 Vertebral Levels
Completed | 20; 55 Vertebral Levels | 20; 55 Vertebral Levels
Not Completed | 1; 3 Vertebral Levels | 1; 3 Vertebral Levels
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Study Arm: Participants will be entered into the single armed study in which one side of the fusion will be coated with milled local autograft bone and the opposite fusion side will be supplemented with an equal volume of Depuy Synthes ViviGen.
  ViviGen Cellular Bone Matrix: Study participants will receive local autograft milled bone on one side of the fusion and an equal amount of Depuy Synthes ViviGen on the opposite side of the fusion
Arm/Group | Study Arm
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.95 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: The Number of Surgical Levels With Successful Lumbar Fusion
Description: Extent of fusion using the Lenke classification. Radiographic success defined as grade A, partial success grade B and radiographic failure as grades C and D.
Time Frame: 12 months prospective from surgery
Population: Surgical Levels have two sides being evaluated: 55 levels times 2: (Left- Autograft and Right - ViviGen)
Measure: Number; unit: Surgical Levels
Units Other Than Participants: Surgical Levels and Sides
Groups:
- Left Side - Milled Local Autograft Bone: Left side of the fusion will be coated with milled local autograft bone.
- Right Side - Depuy Synthes ViviGen: The Right fusion side will be supplemented with Depuy Synthes ViviGen.
Arm/Group | Left Side - Milled Local Autograft Bone | Right Side - Depuy Synthes ViviGen
Number analyzed (Participants) | 20 | 20
Number analyzed (Surgical Levels and Sides) | 55 | 55
Surgical Levels
  Grade A | 24 | 34
  Grade B | 14 | 9
  Grade C | 15 | 12
  Grade D | 2 | 0

2. Secondary Outcome: Number of Participants With or Without Changes in Visual Analog Scale Pain Scores
Description: The visual analog scale will be used to rate leg and back pain scores from 0-10, with 10 being considered the most painful.
Time Frame: 12 months prospectively from surgery
Measure: Number; unit: participants
Arm/Group | Study Arm
Number analyzed (Participants) | 20
participants
  Back Pain Scores Improved on Scale | 12
  Leg Pain Scores Improved on Scale | 11
  Back Pain Scores Worsened on Scale | 2
  Leg Pain Score Worsened on Scale | 1
  Back Pain Score did not change | 2
  Leg Pain Score did not change | 3
  Back Pain Change Unknown/Unreported | 4
  Leg Pain Change Unknown/Unreported | 5

3. Secondary Outcome: Oswestry Disability Index (ODI) v2.1a
Description: This survey will be used to assess how back pain affects patients' ability to function in everyday life. We will look to see if subjects' scores improve or worsen on the Oswestry Disability Index scale (ODI) which can range from 0% to 100% with higher scores indicating higher levels of disturbance in everyday life.
Time Frame: 12 months prospectively from surgery
Measure: Number; unit: participants
Arm/Group | Study Arm
Number analyzed (Participants) | 20
participants
  Oswestry Disability Index Score Improved | 9
  Oswestry Disability Index Score Worsened | 3
  Oswestry Disability Index Score did not Change | 1
  Oswestry Disability Index Score Unknown/Not Reported | 7

ADVERSE EVENTS:
Time Frame: Minimum of 1 year (2 years as available).
Arm/Group | Study Arm
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 6/21
Other Adverse Events (participants affected / at risk) | 14/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm (N=21)
Alcohol Withdrawal (General disorders) | 1 (1)
Shoulder Surgeries (Surgical and medical procedures) | 1 (1)
Altered Mental State (Psychiatric disorders) | 1 (1)
Atrial Fibrillation (AFib) With Rapid Ventricular Response (RVR) (Cardiac disorders) | 1 (1)
Hip Arthroplasties (Surgical and medical procedures) | 1 (1)
Wound Dehiscence (Infections and infestations) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
subdural hematoma (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm (N=21)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
Worsened Back and/or Leg Pain (Musculoskeletal and connective tissue disorders) | 3 (4) — New onset of pain. Possibly a result of a fall or injury.
Epigastric or Abdominal Pain (Gastrointestinal disorders) | 3 (3) — Ex: gastritis or hernia
Increased Paresthesia or Weakness (Nervous system disorders) | 5 (5) — Legs and/or back
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) — Post-operative ileus
Falls or injury (General disorders) | 1 (2) — Not resulting in back or leg injury (other).
Viral Infections (Infections and infestations) | 1 (1) — Coronavirus or flu
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal Cell Carcinoma (Skin and subcutaneous tissue disorders) | 1 (1)
New Diagnosis of Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Adjacent Segment Disease (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Primary Investigator left the university leading to early termination with a small number of subjects analyzed in an interim analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/94/NCT04007094/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/94/NCT04007094/ICF_001.pdf